CLINICAL TRIAL: NCT02086786
Title: Multicenter, Open-label, Two-arm, Parallel-design, Repeat-dose Clinical Trial to Evaluate the PK, Safety, and Tolerability of Four Intramuscular Injections of Risperidone ISM® 75 mg, at 28 Day Intervals in Patients With Schizophrenia
Brief Title: Pharmacokinetics and Tolerability Study of Risperidone ISM® in Schizophrenia
Acronym: PRISMA-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rovi Pharmaceuticals Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROV-RISP-2011-02
Record Dates: First submitted 2014-02-10; First posted 2014-03-13 (Estimated); Results first posted 2017-07-13 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2015-05

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gluteus (Risperidone ISM) (Experimental): Risperidone ISM (75 mg) injection in the gluteal muscle at 28-day intervals
  Interventions: Drug: Risperidone ISM
- Deltoid (Risperdione ISM) (Experimental): Risperidone ISM (75 mg) injection in the deltoid muscle at 28-day intervals
  Interventions: Drug: Risperidone ISM

INTERVENTIONS:
Drug: Risperidone ISM — Four doses of 75 mg of Risperidone ISM as intramuscular (IM) injection into the deltoid muscle at 28-day intervals.
  Four doses of 75 mg of Risperidone ISM as intramuscular injections into the gluteal muscle at 28-day intervals.
  Other Names: No other names

SUMMARY:
To characterize the pharmacokinetics (PK) of the injectable intramuscular (IM) long-acting formulation (in situ microparticle, ISM) of risperidone over four IM injections in the gluteal and deltoid muscle at 28-day intervals and at one dose strength (75 mg) in patients with schizophrenia.

DETAILED DESCRIPTION:
This was a multicenter, open-label, two-arm, parallel-design, repeat-dose clinical study designed to evaluate the PK, safety, and tolerability of Risperidone ISM®, a new long-acting injectable formulation of the licensed drug risperidone, administered in the gluteal muscle or the deltoid muscle. Participants were patients with a diagnosis of schizophrenia capable of understanding, signing, and consenting to study participation on their own.

Objectives:

Primary Objective

• To characterize the pharmacokinetics (PK) of the injectable intramuscular (IM) long-acting formulation of risperidone over four IM injections in the gluteal and deltoid muscle at 28 day intervals and at one dose strength (75 mg) in patients with schizophrenia.

Secondary Objectives

* To document the attainment of steady-state exposure by the injectable formulation ISM® of risperidone over four IM injections in the gluteal and deltoid muscle at 28-day intervals and at one dose strength (75 mg) in patients with schizophrenia.
* To perform a descriptive comparison of the PK data between the gluteal and the deltoid muscle administration of the injectable formulation ISM® of risperidone over four IM injections at 28-day intervals and at one dose strength (75 mg) in patients with schizophrenia.
* To evaluate the safety and tolerability of the injectable formulation ISM® of risperidone after four IM injections in the gluteal muscle or deltoid muscle at 28-day intervals at one dose strength (75 mg) in patients with schizophrenia.

Exploratory Objectives

* To explore the efficacy of once every four weeks of the injectable formulation ISM® of risperidone after four IM injections in the gluteal muscle or deltoid muscle at 28-day (± 1 day) intervals at one dose strength (75 mg) in patients with schizophrenia.
* To characterize patients' metabolic phenotype (cytochrome P450 [CYP]2D6, CYP3A4) to explain any potential unexpected outlying PK value, and/or explore its relationship with any potential safety or tolerability issue.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of providing informed consent.
2. Male or female aged ≥18 years to ≤65 years.
3. Current diagnosis of schizophrenia, according to Diagnostic and Statistical Manual
4. Body mass index (BMI) ≥17 kg/m2 but ≤35 kg/m2.
5. Medically stable over the last month, and psychiatrically stable
6. On oral stable dosage of risperidone ≥4 mg daily as maintenance therapy.
7. Total score ≤70 on the Positive and Negative Syndrome Scale.
8. Using a medically accepted contraceptive method
9. Agrees to washout all prohibited medications prior to baseline (day -1)

Exclusion Criteria:

1. Informed consent obtained from a third party.
2. Prisoners or patients who are compulsorily detained.
3. Females who are breast-feeding and/or who have a positive pregnancy test.
4. Presence of an uncontrolled, unstable clinically significant medical condition.
5. Positive serology for Hepatitis B, Hepatitis C or anti-HIV 1 and 2 at screening.
6. History of neuroleptic malignant syndrome.
7. Current or past history of tardive dyskinesia.
8. Positive urine drug or alcohol screen finding.
9. Risk of committing self-harm or harm based on Columbia Suicidal Rating Scale.
10. Taking more than one antidepressant.
11. Use of depot antipsychotics within the last three months.
12. Use of strong or moderate cytochrome P450 isoenzyme 3A4inducers
13. Use of electroconvulsive therapy (ECT) within the last three months.
14. Receipt of any investigational drugs within the last three months.
15. Known or suspected allergy or hypersensitivity to risperidone
16. Previous non-responder to risperidone treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Llaudó, M.D, Study Chair — Rovi Laboratorios Farmacéuticos
Locations (1):
- St Louis Clinical Trials, LC, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Gluteus (Risperidone ISM): Risperidone ISM (75 mg) injection in the gluteal muscle at 28-day intervals
  Risperidone ISM
- Deltoid (Risperdione ISM): Risperidone ISM (75 mg) injection in the deltoid muscle at 28-day intervals
  Risperidone ISM
Period: Overall Study
Arm/Group | Gluteus (Risperidone ISM) | Deltoid (Risperdione ISM)
Started | 35 | 35
Completed | 17 | 19
Not Completed | 18 | 16

BASELINE CHARACTERISTICS:
Population: Three of the randomized patients (70) were not dosed. Two of them due to withdrawal of consent and the third due to fulfilment of one of the study exclusion criteria (take prohibited medication). Thus, the number of patients receiving the study medication were 67; 34 in the gluteal injection group and 33 in the deltoid injection group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Gluteus (Risperidone ISM) | Deltoid (Risperdione ISM) | Total
Number analyzed (Participants) | 34 | 33 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 33 | 67
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (11.1) | 44 (9.8) | 43 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 27 | 28 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 28 | 53
  White | 7 | 4 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 33 | 67

OUTCOME MEASURES:

1. Primary Outcome: Peak Plasma Concentration (Cmax) for Active Moiety
Time Frame: Dose 1, 2 and 3: Pre-dose; at 2, 8, 12, 24 and 48 hours post-dose; 5, 7, 10, 14, 18, and 21 days post-dose. Dose 4: Pre dose; at 2, 8, 12, 24, and 48 hours post-dose; at 5, 7, 10, 14, 18, 21, 25, 28, 32, 37, 42, 60, 75, 90, 105, and 120 days post-dose.
Population: The analysis was conducted in the PK population, which includes 43 patients (20 in the gluteal and 23 in the deltoid site injection group) who had at least 1 PK sample taken and had no major protocol deviations that would exclude them from PK analysis. They also had concentration data amenable to evaluation as determined by the pharmacokineticist.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Gluteus (Risperidone ISM): Risperidone ISM (75 mg) injection in the gluteal muscle at 28-day intervals
  Risperidone ISM: Four doses of 75 mg of Risperidone ISM as intramuscular (IM) injection into the deltoid muscle at 28-day intervals.
  Four doses of 75 mg of Risperidone ISM as intramuscular injections into the gluteal muscle at 28-day intervals.
- Deltoid (Risperdione ISM): Risperidone ISM (75 mg) injection in the deltoid muscle at 28-day intervals
  Risperidone ISM: Four doses of 75 mg of Risperidone ISM as intramuscular (IM) injection into the deltoid muscle at 28-day intervals.
  Four doses of 75 mg of Risperidone ISM as intramuscular injections into the gluteal muscle at 28-day intervals.
Arm/Group | Gluteus (Risperidone ISM) | Deltoid (Risperdione ISM)
Number analyzed (Participants) | 20 | 23
ng/mL
  Dose 1 | 39.6 (33.7) | 54.1 (48.9)
  Dose 2 | 53.2 (52.7) | 61.0 (38.4)
  Dose 3 | 48.6 (33.3) | 61.0 (36.9)
  Dose 4 | 47.4 (38.9) | 57.7 (39.3)

2. Primary Outcome: Trough Plasma Concentration (Cmin) for Active Moiety
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Gluteus (Risperidone ISM) | Deltoid (Risperdione ISM)
Number analyzed (Participants) | 20 | 23
ng/mL
  Dose 1 | 11.1 (72.6) | 7.0 (87.6)
  Dose 2 | 7.86 (90.1) | 8.60 (49.4)
  Dose 3 | 9.97 (70.7) | 10.2 (57.6)
  Dose 4 | 12.6 (59.1) | 9.52 (56.5)

3. Primary Outcome: Area Under the Curve to the Last Quantified Concentration (AUClast) for Active Moiety
Time Frame: as for outcome 1
Population: The analysis was conducted in the PK population (patients who had at least 1 PK sample taken and had no major protocol deviations that would exclude them from PK analysis). As determined by the pharmacokineticist, for this analysis, 18 patients in the gluteal and 22 in the deltoids had concentration amenable to evaluation..
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Gluteus (Risperidone ISM) | Deltoid (Risperdione ISM)
Number analyzed (Participants) | 18 | 22
h*ng/mL | 21300 (35.2) | 23300 (43.3)

4. Primary Outcome: Area Under the Curve Extrapolated to Infinity (AUC∞) for Active Moiety
Time Frame: as for outcome 1
Population: The analysis was conducted in the PK population (patients who had at least 1 PK sample taken and had no major protocol deviations that would exclude them from PK analysis). As determined by the pharmacokineticist, for this analysis, 11 patients in the gluteal and 18 in the deltoids had concentration amenable to evaluation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Gluteus (Risperidone ISM) | Deltoid (Risperdione ISM)
Number analyzed (Participants) | 11 | 18
h*ng/mL | 21100 (27.4) | 22700 (40.4)

5. Primary Outcome: AUCτ for Active Moiety
Description: AUCτ is the area under the curve over the dosing interval (τ), where the dosing interval is 28 days
Time Frame: as for outcome 1
Population: The analysis was conducted in the PK population: 43 patients (20 in the gluteal and 23 in the deltoid site injection group). As determined by the pharmacokineticist, for Dose 4th analysis, 18 patients in the gluteal and 22 in the deltoid group had concentration amenable to evaluation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Gluteus (Risperidone ISM) | Deltoid (Risperdione ISM)
Number analyzed (Participants) | 20 | 23
h*ng/mL
  Dose 1 | 14100 (39.5) | 16300 (42.6)
  Dose 2 | 15400 (59.3) | 18000 (40.2)
  Dose 3 | 16600 (24.2) | 18200 (32.5)
  Dose 4 | 17300 (27.1) | 18500 (35.9)

6. Primary Outcome: Time to Peak Concentration (Tmax) for Active Moiety
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | Gluteus (Risperidone ISM) | Deltoid (Risperdione ISM)
Number analyzed (Participants) | 20 | 23
h
  Dose 1 | 48.0 [23.9 to 504] | 48.0 [23.8 to 216]
  Dose 2 | 24.0 [2.0 to 48.1] | 24.0 [2.08 to 479]
  Dose 3 | 48.0 [12.0 to 504] | 24.0 [2.0 to 215]
  Dose 4 | 24.0 [7.97 to 502] | 48.0 [2.13 to 505]

7. Primary Outcome: Terminal Half-life (t1/2) for Active Moiety
Time Frame: as for outcome 1
Population: The analysis was conducted in the PK population (patients who had at least 1 PK sample taken and had no major protocol deviations that would exclude them from PK analysis). As determined by the pharmacokineticist, for this analysis, 12 patients in the gluteal and 19 in the deltoid group had concentration amenable to evaluation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Gluteus (Risperidone ISM) | Deltoid (Risperdione ISM)
Number analyzed (Participants) | 12 | 19
h | 163 (80.5) | 269 (71.6)

8. Primary Outcome: PTF for Active Moiety
Description: Peak to Trough Fluctuation ratio for the Active Moiety
Time Frame: as for outcome 1
Population: The analysis was conduct in the PK population, which includes 43 patients (20 in the gluteal and 23 in the deltoid site injection group) who had at least 1 PK sample taken and had no major protocol deviations that would exclude them from PK analysis. They also had concentration data amenable to evaluation as determined by the pharmacokineticist.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Gluteus (Risperidone ISM) | Deltoid (Risperdione ISM)
Number analyzed (Participants) | 20 | 23
Ratio
  Dose 1 | 0.999 (181.6) | 1.76 (47.6)
  Dose 2 | 1.89 (38.1) | 1.88 (23.0)
  Dose 3 | 1.39 (51.9) | 1.82 (29.6)

9. Secondary Outcome: Accumulation Ratio (RA) for Active Moiety
Description: Defined as AUC (0-28 days) after the 4th dose divided by the AUC (0-28 days) of the first dose.
Time Frame: as for outcome 1
Population: The analysis was conducted in the PK population (patients who had at least 1 PK sample taken and had no major protocol deviations that would exclude them from PK analysis). As determined by the pharmacokineticist, for this analysis, 18 patients in the gluteal and 22 in the deltoid group had concentration amenable to evaluation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Gluteus (Risperidone ISM) | Deltoid (Risperdione ISM)
Number analyzed (Participants) | 18 | 22
Ratio | 1.15 (25.1) | 1.14 (26.2)

10. Other Pre Specified Outcome: Positive and Negative Syndrome Scale (PANSS) Total Score
Description: The change in PANSS score from Baseline by visit 48.
  The PANSS combines 3 subscales: The positive scale (7 items), the negative scale (7 items) and the general psychopathology scale (16 items).
  PANSS Items Scores: 1 = Absent, 2 = Minimal, 3 = Mild, 4 = Moderate, 5 = Moderate Severe, 6 = Severe, 7 = Extreme.
  Subscales are summed to compute a total score Range for each of the subscales: Positive scale (7-49); Negative scale (7-49); General psychopathology scale (16-112) Range for the PANSS total scale: 30-210 PANSS total score ≤70: stable schizophrenia PANSS total score between >70: decompensated schizophrenia
Time Frame: Baseline, Days 5, 7, 10, 14, 18, and 21 post Dose 1; Dose 2, 3 and 4 post dose; Days 5, 7, 10, 14, 18, and 21 post Dose 2, 3, and 4; Days 25, 28, 32, 37, 42, 60, 75, 90, and 105 post Dose 4; Day 120 post Dose 4 or early termination.
Population: The analysis was conduct in the Intent-to-Treat (ITT) Population, which includes all patients in Safety Population with baseline (Day -1) efficacy data and at least 1 post-baseline efficacy evaluation. ITT Population includes 66 patients; 33 on each arm.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Gluteus (Risperidone ISM) | Deltoid (Risperdione ISM)
Number analyzed (Participants) | 33 | 33
points
  Baseline (Day -1) | 58 (10.4) | 60 (9.8)
  Visit 48 (Day 120 post Dose 4) | 59 (16.4) | 61 (10.8)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected in all visits of the study: Screening, Baseline (Day -1); Day 0 (Dose 1); Days 1, 2, 5, 7, 10, 14, 18 & 21 Post Dose 1; Dose 2, 3 & 4 Prior to Dosage and Post Dose; Days 1, 2, 5, 7, 10, 14, 18 & 21 Post Dose 2, 3 & 4; Days 25, 28, 32, 37, 42, 60, 75, 90 & 105 Post-Dose 4; Day 120 Post-Dose 4 (final visit) or any Early Termination.
Description: The analysis was performed in the Safety Population, which includes all patients who received at least 1 dose of the study drug: 67 patients in total, 34 of them were in the gluteal arm and 33 in the Deltoid arm. This is the population at risk.
Arm/Group | Gluteus (Risperidone ISM) | Deltoid (Risperdione ISM)
Serious Adverse Events (participants affected / at risk) | 5/34 | 7/33
Other Adverse Events (participants affected / at risk) | 32/34 | 31/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gluteus (Risperidone ISM) (N=34) | Deltoid (Risperdione ISM) (N=33)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oromandibular dystonia (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Drug abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Schizophrenia (Psychiatric disorders) | 0 (0) | 3 (3)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gluteus (Risperidone ISM) (N=34) | Deltoid (Risperdione ISM) (N=33)
Hyperprolactinaemia (Endocrine disorders) | 19 (55) | 17 (41)
Tachycardi (Cardiac disorders) | 0 (0) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (3)
Fatigue (General disorders) | 1 (1) | 2 (2)
Injection site erythema (General disorders) | 7 (12) | 3 (6)
Injection site induration (General disorders) | 1 (2) | 4 (4)
Injection site pain (General disorders) | 12 (31) | 10 (25)
Pain (General disorders) | 3 (4) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
ECG QT prolonged (Investigations) | 0 (0) | 2 (3)
Heart rate increased (Investigations) | 1 (1) | 2 (2)
Muskuloskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Akathisia (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 4 (4) | 2 (2)
Drooling (Nervous system disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 4 (7) | 1 (1)
Oromandibular dystonia (Nervous system disorders) | 2 (2) | 7 (8)
Sedation (Nervous system disorders) | 6 (7) | 4 (5)
Somnolence (Nervous system disorders) | 2 (2) | 7 (8)
Schizophrenia (Psychiatric disorders) | 2 (2) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor intends to publish clinical data from all centers participating in the investigation. A draft manuscripts will submit to all participating investigators for their comments. Individual investigators subsequently may publish additional findings of this study in scientific journals/scientific meetings, provided that the sponsor is given ample opportunity to review any proposed abstract, manuscript, or slide presentation prior to its submission.